CLINICAL TRIAL: NCT05664906
Title: Evaluating Efficacy and Safety of Chinese Medicine Oral Rinse in Treating and Preventing Irradiated Oral Mucositis in Head-and-Neck Cancer Patients - a Pilot Trial
Brief Title: Evaluating Chinese Medicine Oral Rinse for Irradiated Oral Mucositis in Head & Neck Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Au Kwok Yin, Dr. AU Kwok Yin, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM Rinse_OMRT
Record Dates: First submitted 2022-11-06; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Neoplasms; Oral Mucositis (Ulcerative) Due to Radiation; Chinese Medicine Oral Rinse
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A randomized controlled pilot study will be employed, participants will receive either CM Oral Rinse granules (CMORF-I) or placebo while they will receive standard care too. Since the duration of RT and recruitment time may vary, the intervention period starts from baseline (14 days within RT starts) to 2 weeks after the end of RT, while the post-intervention period will be 10 weeks starting from 2 weeks after the end of RT with 3 post-intervention follow-up visits (4 weeks, 8 weeks and 12 weeks after the end of RT).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Chinese Medicine Oral Rinse and Standard Care (Active Comparator): * Prescription and oral rinsing with Chinese Medicine Oral Rinse Formula-I (CMORF-I) which mainly consists of the Nong's concentrated CM granules of Wu Wei Xiao Du Yin and other ingredients.
  * Standard care will be following the indications provided by patient's western medical doctor.
  * Patients should not take any other TCM and non-prescribed medication and nutritional supplements during the intervention period.
  Interventions: Drug: Chinese Medicine Oral Rinse Formula-I (CMORF-I); Other: Standard Care
- Control Group: Placebo and Standard Care (Placebo Comparator): * Placebo: The placebo consists of an inert substance, made of starch filler, flavor and colorings. It is also manufactured under GMP standard. To ensure blinding, the CMORF-I formula and placebo will be indistinguishable in appearance, smell and favour.
  * Standard care will be following the indications provided by patient's western medical doctor.
  * Patients should not take any other TCM and non-prescribed medication and nutritional supplements during the intervention period.
  Interventions: Other: Standard Care; Other: Placebo

INTERVENTIONS:
Drug: Chinese Medicine Oral Rinse Formula-I (CMORF-I) — * Prescription of Chinese Medicine Oral Rinse Formula-I (CMORF-I)
  * Instruction to rinse:
    1. The above amount of concentrated CM granules will be divided and packed in 4 bags per day.
    2. Dissolve 1 bag of concentrated CM granules with 150ml 80'C boiled hot water, and wait for 20 mins to cool down.
    3. Clean the mouth thoughtfully by rinsing with 150ml of distilled water for 2 minutes.
    4. Rinse the mouth thoughtfully with one-third of the dissolved and cooled CM oral rinse, gargle, expel after 3 minutes, do not swallow and repeat twice.
    5. To ensure better contact of the CM oral rinse in all parts and folds of the oral cavity, our research assistant and CMP will guide the patients to fully agitate the mouth, use the tongue to stir repeatedly among the teeth, cheeks and palate surface, and to raise the tip of the tongue for a moment and tilt the head back.
    6. 4 times a day (half an hour after every meal, half an hour before sleep), from baseline to 2 weeks after RT.
  Other Names: CMORF-I
  Arms: Intervention Group: Chinese Medicine Oral Rinse and Standard Care
Other: Standard Care — • Standard care including normal saline or medical mouthwash, optional analgesics and antibiotics will be offered by hospital.
Other: Placebo — Placebo granules, instruction is the same as CMORF-I.
  Arms: Control Group: Placebo and Standard Care

SUMMARY:
Approximately 60% and 90% of patients with head and neck (H&N) cancers receiving standard radiotherapy (RT) and chemoradiotherapy (chemo-RT) will develop oral mucositis respectively. Oral mucositis (OM) is one of the dose-limiting adverse events which can also lead to emotional and nutritional problems. Clinically, it is usually observed by the end of first week of RT (after 10 Gy) and reaches peak damage in 14-21 days or by the end of treatment. Healing then takes approximately 2 to 3 weeks after completion of RT. For the Chinese Medicine (CM) interventions, many studies have been reviewed on the efficacy of mouthwash or internal herbal decoction to OM. Although some positive results were observed, most of them were performed by applying different assessment tools and lack of quality of life (QOL) or self-reported symptoms assessment. In addition, the intervention time and follow-up period were usually insufficient (stopped at the end of RT), therefore they could not review the long-term efficacy of CM according to normal progression of OM and the safety of using CM. Therefore, we hope this pilot study can evaluate the efficacy and safety of CM in a strict protocol.

DETAILED DESCRIPTION:
Approximately 60% and 90% of patients with head and neck (H&N) cancers receiving standard radiotherapy (RT) and chemoradiotherapy (chemo-RT) will develop oral mucositis respectively. Oral mucositis (OM) is one of the dose-limiting adverse events which can also lead to emotional and nutritional problems. Clinically, it is usually observed by the end of first week of RT (after 10 Gy) and reaches peak damage in 14-21 days or by the end of treatment. Healing then takes approximately 2 to 3 weeks after completion of RT.

The risk of OM is especially high in NPC patients who receive concomitant chemotherapy, receive a total dose over 5,000 Gy, treat with altered fractionation radiation schedules, have bad oral hygiene status, do not use antibiotic at early stage mucositis, have smoking history, drink alcohol, have problems in nutritional status like anorexia, malnutrition, lack of vitamins, restriction of food due to specific dietary requirements, have haematological disease or non-ideal hematological status, have advanced localization of tumors and stage, receive immunotherapy, have pre-existing dry mouth (Xerostomia), have episodes of OM during prior treatment cycles and low BMI, etc.

According to some weighed guidelines such as The Multinational Association of Supportive Care in Cancer and International Society for Oral Oncology (MASCC/ISOO) guidelines for the management of OM, recent systematic reviews and researches, there are mainly several sections for intervention: (1) Basic oral care, (2) Anti-inflammatory agents, (3) Photobiomodulation, (4) Cryotherapy, (5) Antimicrobials, coating agents, anesthetics, and analgesics, (6) Growth factors and cytokines, and (7) Natural and miscellaneous. We can summarize several suggestions for the prevention of OM in H&N cancer adults receiving RT from the above protocols: multiagent combination oral care protocols (increasing the awareness of good oral hygiene), professional dental care (a desirable option before or during cancer therapy for local and systemic infections from odontogenic sources), benzydamine mouthwash (as the anti-inflammaotary agents for moderate dose of RT (<50 Gy)) and intraoral photobiomodulation therapy using low-level laser therapy. Over the years, the number of interventions studied for OM and their quality of study design have been dramatically increasing. However, since there are still some advantages and disadvantages for some suggested agents, some clinical settings have not yet been recommended with appropriate intervention. Natural and miscellaneous agents are also reviewed in the past years while honey is suggested for prevention of OM in patients with H&N cancer who receive treatment with either RT or chemo-RT. However, if honey is applied repeatedly on a daily basis for a longer period, we have to be cautions with its deleterious effects. A strict oral hygiene protocol has to be followed to prevent dental caries.

For the Chinese Medicine (CM) interventions, many studies have been reviewed on the efficacy of mouthwash or internal herbal decoction to OM. Although some positive results were observed, most of them were performed by applying different assessment tools and lack of quality of life (QOL) or self-reported symptoms assessment. In addition, the intervention time and follow-up period were usually insufficient (stopped at the end of RT), therefore they could not review the long-term efficacy of CM according to normal progression of OM and the safety of using CM. Therefore, we hope this pilot study can evaluate the efficacy and safety of CM in a strict protocol.

ELIGIBILITY:
Inclusion Criteria: Patients who

* are aged ≥18, with known diagnosis of non-metastatic hypopharyngeal cancer, laryngeal cancer, lip and oral cavity cancer, nasopharyngeal cancer, oropharyngeal cancer, paranasal sinus and nasal cavity cancer, and salivary gland cancer.
* are the first time to receive RT to the primary tumor in the area of the head or face, neck, or oral cavity.
* start RT recently within 14 days.
* are assessed by CMPs for the condition of oral mucositis according to modified World Health Organization (WHO) Mucositis Grades with Grade ≦1.
* have Karnofsky Performance Status (KPS) ≥ 60 (patients require occasional assistance, but is able to care for most personal needs will be 60 or above).
* are able to read or understand and sign the consent form.

Exclusion Criteria: Patients who

* receive concurrent chemo-radiation.
* have known medication on bacterial or fungal infections of oropharynx at recruitment.
* have other known diseases such as serious and uncontrolled Diabetes mellitus (with symptom of delayed wound healing over the past half year) or hyperthyroidism (with symptom of serious oral dryness over the past half year), known connective vascular disorders or known Human Immunodeficiency Virus (HIV) infections etc.
* have known history of allergy to CMORF-I ingredients or Glucose-6-Phosphate Dehydrogenase (G6PD) patients.
* are known pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of the most severe modified WHO Mucositis Grades | From baseline to week 12 after the end of RT during post intervention period
  * Comparison of the proportion of the most severe modified WHO Mucositis Grades among intervention and control groups during RT.
  * Grades of the OM will be assessed by a Registered Chinese medicine practitioner (CMP) at baseline and day 7 (±1d) of every week during the RT, the most severe grades during the treatment will be regarded for data analysis.
  * Modified WHO Mucositis Grading Scale: Grade 0 (none) - normal; Grade 1 (mild) - soreness/erythema; Grade 2 (moderate) - erythema, ulcer/pseudo-membranes, can eat solids (erythema with ulcers less than 1 cm); Grade 3 (severe) - ulcer/pseudo-membrane, (erythema with ulcers more than 1cm) requires liquid diet only; Grade 4 (life-threatening) - ulcer with hemorrhage and necrosis, alimentation not possible; cancer treatment that results in or contribute to death is reported separately.

SECONDARY OUTCOMES:
10cm visual analogue scale (VAS) of oral pain | Day 3 and day 7 (±1d) of every week during intervention period, end of week 4, week 8 and week 12 after the end of RT during post intervention period.
  It is a measurement of oral pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" on the left and "worst pain" on the right.
Oral Mucositis Daily Questionnaire (OMDQ) (validated Chinese version with modification) | Day 3 and day 7 (±1d) of every week during intervention period, once a week during post intervention period, end of week 4, week 8 and week 12 after the end of RT during post intervention period.
  It is a measurement of self-reported quality of life. It contains 10 items, for most questions in the OMDQ, a higher score indicated a worsening in symptom severity or more interference with functional activity. For the question pertaining to overall health, a higher score indicates better overall health status.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (Head and Neck) (EORTC QLQ-C30) (Hong Kong Cantonese version) | Day 7 (±1d) of every week during intervention period, end of week 4, week 8 and week 12 after the end of RT during post intervention period.
  It is a specific measurement of self-reported quality of life for Head and Neck cancer patients. It consists of 30 questions that indicate the extent to which you have experienced these symptoms or problems during the past week. Scoring from 1 "Not at all" to 4 "Very much".
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (Head and Neck) (EORTC QLQ-H&N35) (Hong Kong Cantonese version) | Day 7 (±1d) of every week during intervention period, end of week 4, week 8 and week 12 after the end of RT during post intervention period.
  It is a specific measurement of self-reported quality of life for Head and Neck cancer patients. It consists of 35 questions that indicate the extent to which you have experienced these symptoms or problems during the past week. Scoring from 1 "Not at all" to 4 "Very much".
Body mass index (BMI) | From baseline to week 12 after the end of RT during post intervention period
  It is a measurement of the amount of body fat based on height and weight that applies to adult men and women. It can assess and monitor the risk of OM to a certain extent.
Number of analgesic and antibiotics use daily | From baseline to week 12 after the end of RT during post intervention period
  It can assess and monitor the conditions of OM.

CONTACTS AND LOCATIONS:
Overall Officials: KWOK YIN AU, Doctor of Medicine, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- Hong Kong Institute of Integrative Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. WHO Handbook for Reporting the Results of Cancer Treatment. Geneva: WHO Offset Publications, 1979; 48:15-22
- [Background] National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE 4.03) from: https://ctep.cancer.gov/protocolDevelopment/adverse_effects.htm
- [Background] Chinese Pharmacopoeia Commission. Pharmacopoeia of the People's Republic of China (English Edition) Vol. 1. Beijing, China: China Medical Science Press; 2015.
- [Result] Sutherland SE, Browman GP. Prophylaxis of oral mucositis in irradiated head-and-neck cancer patients: a proposed classification scheme of interventions and meta-analysis of randomized controlled trials. Int J Radiat Oncol Biol Phys. 2001 Mar 15;49(4):917-30. doi: 10.1016/s0360-3016(00)01456-5. PMID 11240232
- [Result] Lichtman SM. Physiological aspects of aging. Implications for the treatment of cancer. Drugs Aging. 1995 Sep;7(3):212-25. doi: 10.2165/00002512-199507030-00006. PMID 8535051
- [Result] Ps SK, Balan A, Sankar A, Bose T. Radiation induced oral mucositis. Indian J Palliat Care. 2009 Jul;15(2):95-102. doi: 10.4103/0973-1075.58452. PMID 20668585
- [Result] Luo DH, Hong MH, Guo L, Cao KJ, Deng MQ, Mo HY. [Analysis of oral mucositis risk factors during radiotherapy for nasopharyngeal carcinoma patients and establishment of a discriminant model]. Ai Zheng. 2005 Jul;24(7):850-4. Chinese. PMID 16004814
- [Result] Saito N, Imai Y, Muto T, Sairenchi T. Low body mass index as a risk factor of moderate to severe oral mucositis in oral cancer patients with radiotherapy. Support Care Cancer. 2012 Dec;20(12):3373-7. doi: 10.1007/s00520-012-1620-7. Epub 2012 Oct 7. PMID 23052923
- [Result] Elad S, Cheng KKF, Lalla RV, Yarom N, Hong C, Logan RM, Bowen J, Gibson R, Saunders DP, Zadik Y, Ariyawardana A, Correa ME, Ranna V, Bossi P; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2020 Oct 1;126(19):4423-4431. doi: 10.1002/cncr.33100. Epub 2020 Jul 28. PMID 32786044
- [Result] Rashad UM, Al-Gezawy SM, El-Gezawy E, Azzaz AN. Honey as topical prophylaxis against radiochemotherapy-induced mucositis in head and neck cancer. J Laryngol Otol. 2009 Feb;123(2):223-8. doi: 10.1017/S0022215108002478. Epub 2008 May 19. PMID 18485252
- [Result] Yarom N, Hovan A, Bossi P, Ariyawardana A, Jensen SB, Gobbo M, Saca-Hazboun H, Kandwal A, Majorana A, Ottaviani G, Pentenero M, Nasr NM, Rouleau T, Lucas AS, Treister NS, Zur E, Ranna V, Vaddi A, Barasch A, Lalla RV, Cheng KKF, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer / International Society of Oral Oncology (MASCC/ISOO). Systematic review of natural and miscellaneous agents, for the management of oral mucositis in cancer patients and clinical practice guidelines - part 2: honey, herbal compounds, saliva stimulants, probiotics, and miscellaneous agents. Support Care Cancer. 2020 May;28(5):2457-2472. doi: 10.1007/s00520-019-05256-4. Epub 2020 Feb 13. PMID 32056010
- [Result] Elting LS, Keefe DM, Sonis ST, Garden AS, Spijkervet FK, Barasch A, Tishler RB, Canty TP, Kudrimoti MK, Vera-Llonch M; Burden of Illness Head and Neck Writing Committee. Patient-reported measurements of oral mucositis in head and neck cancer patients treated with radiotherapy with or without chemotherapy: demonstration of increased frequency, severity, resistance to palliation, and impact on quality of life. Cancer. 2008 Nov 15;113(10):2704-13. doi: 10.1002/cncr.23898. PMID 18973181
- [Result] Stiff PJ, Erder H, Bensinger WI, Emmanouilides C, Gentile T, Isitt J, Lu ZJ, Spielberger R. Reliability and validity of a patient self-administered daily questionnaire to assess impact of oral mucositis (OM) on pain and daily functioning in patients undergoing autologous hematopoietic stem cell transplantation (HSCT). Bone Marrow Transplant. 2006 Feb;37(4):393-401. doi: 10.1038/sj.bmt.1705250. PMID 16415901
- [Result] GU, Y., GONG, L., & Yan, H. (2014). Reliability and validity of Chinese version of Oral Mucositis Daily Questionnaire (OMDQ). Chinese Journal of Nursing, 49(1), 108-112.
- [Result] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Result] Stokman MA, Burlage FR, Spijkervet FK. The effect of a calcium phosphate mouth rinse on (chemo) radiation induced oral mucositis in head and neck cancer patients: a prospective study. Int J Dent Hyg. 2012 Aug;10(3):175-80. doi: 10.1111/j.1601-5037.2012.00574.x. PMID 23046006
- [Result] Roopashri G, Jayanthi K, Guruprasad R. Efficacy of benzydamine hydrochloride, chlorhexidine, and povidone iodine in the treatment of oral mucositis among patients undergoing radiotherapy in head and neck malignancies: A drug trail. Contemp Clin Dent. 2011 Jan;2(1):8-12. doi: 10.4103/0976-237X.79292. PMID 22114446
- [Result] Shang X, Pan H, Li M, Miao X, Ding H. Lonicera japonica Thunb.: ethnopharmacology, phytochemistry and pharmacology of an important traditional Chinese medicine. J Ethnopharmacol. 2011 Oct 31;138(1):1-21. doi: 10.1016/j.jep.2011.08.016. Epub 2011 Aug 16. PMID 21864666
- [Result] Li Y, Li W, Fu C, Song Y, Fu Q. Lonicerae japonicae flos and Lonicerae flos: a systematic review of ethnopharmacology, phytochemistry and pharmacology. Phytochem Rev. 2020;19(1):1-61. doi: 10.1007/s11101-019-09655-7. Epub 2019 Nov 22. PMID 32206048
- [Result] Li Y, Cai W, Weng X, Li Q, Wang Y, Chen Y, Zhang W, Yang Q, Guo Y, Zhu X, Wang H. Lonicerae Japonicae Flos and Lonicerae Flos: A Systematic Pharmacology Review. Evid Based Complement Alternat Med. 2015;2015:905063. doi: 10.1155/2015/905063. Epub 2015 Jul 16. PMID 26257818
- [Result] Sun S, Jiang P, Su W, Xiang Y, Li J, Zeng L, Yang S. Wild chrysanthemum extract prevents UVB radiation-induced acute cell death and photoaging. Cytotechnology. 2016 Mar;68(2):229-40. doi: 10.1007/s10616-014-9773-5. Epub 2014 Jul 23. PMID 25052044
- [Result] Luyen BT, Tai BH, Thao NP, Cha JY, Lee HY, Lee YM, Kim YH. Anti-inflammatory components of Chrysanthemum indicum flowers. Bioorg Med Chem Lett. 2015 Jan 15;25(2):266-9. doi: 10.1016/j.bmcl.2014.11.054. Epub 2014 Nov 27. PMID 25497988
- [Result] Shao Y, Sun Y, Li D, Chen Y. Chrysanthemum indicum L.: A Comprehensive Review of its Botany, Phytochemistry and Pharmacology. Am J Chin Med. 2020;48(4):871-897. doi: 10.1142/S0192415X20500421. Epub 2020 May 20. PMID 32431180
- [Result] Hwang ES, Kim GH. Safety Evaluation of Chrysanthemum indicum L. Flower Oil by Assessing Acute Oral Toxicity, Micronucleus Abnormalities, and Mutagenicity. Prev Nutr Food Sci. 2013 Jun;18(2):111-6. doi: 10.3746/pnf.2013.18.2.111. PMID 24471119
- [Result] Schutz K, Carle R, Schieber A. Taraxacum--a review on its phytochemical and pharmacological profile. J Ethnopharmacol. 2006 Oct 11;107(3):313-23. doi: 10.1016/j.jep.2006.07.021. Epub 2006 Jul 22. PMID 16950583
- [Result] Martinez M, Poirrier P, Chamy R, Prufer D, Schulze-Gronover C, Jorquera L, Ruiz G. Taraxacum officinale and related species-An ethnopharmacological review and its potential as a commercial medicinal plant. J Ethnopharmacol. 2015 Jul 1;169:244-62. doi: 10.1016/j.jep.2015.03.067. Epub 2015 Apr 6. PMID 25858507
- [Result] Du D, Cheng Z, Chen D. Anti-complement sesquiterpenes from Viola yedoensis. Fitoterapia. 2015 Mar;101:73-9. doi: 10.1016/j.fitote.2014.12.015. Epub 2015 Jan 3. PMID 25562805
- [Result] Xie C, Kokubun T, Houghton PJ, Simmonds MS. Antibacterial activity of the Chinese traditional medicine, Zi Hua Di Ding. Phytother Res. 2004 Jun;18(6):497-500. doi: 10.1002/ptr.1497. PMID 15287078
- [Result] Jeong YH, Oh YC, Cho WK, Shin H, Lee KY, Ma JY. Anti-inflammatory effects of Viola yedoensis and the application of cell extraction methods for investigating bioactive constituents in macrophages. BMC Complement Altern Med. 2016 Jun 14;16:180. doi: 10.1186/s12906-016-1142-9. PMID 27301877
- [Result] Su Y, Zhang Z, Guo C. A new nitroethylphenolic glycoside from Semiaquilegia adoxoides. Fitoterapia. 2004 Jun;75(3-4):420-2. doi: 10.1016/j.fitote.2004.01.016. PMID 15159012
- [Result] Yang Y, Guo L, Tariq K, Zhang W, Li C, Memon FQ, Chai B, Li Z, Sun J, Chen Y, Zhang G, Li Q, Wang S, Wang L, Lai C, Jiang M, Si H. The Antioxidant Polysaccharide from Semiaquilegia adoxoides (DC.) Makino Adjusts the Immune Response of Mice Infected by Bacteria. Evid Based Complement Alternat Med. 2020 Feb 19;2020:2719483. doi: 10.1155/2020/2719483. eCollection 2020. PMID 32148535
- [Result] Duan SP, Jin CL, Hao J, Hou LJ, Li AH, Zhu ZP, Gao JH, Pan Y. A study on the inhibitory effect of Radix Semiaquilegiae extract on human hepatoma HEPG-2 and SMMC-7721 cells. Afr J Tradit Complement Altern Med. 2013 Aug 12;10(5):336-40. doi: 10.4314/ajtcam.v10i5.19. eCollection 2013. PMID 24311846
- [Result] Jiang F, Li W, Huang Y, Chen Y, Jin B, Chen N, Ding Z, Ding X. Antioxidant, antityrosinase and antitumor activity comparison: the potential utilization of fibrous root part of Bletilla striata (Thunb.) Reichb.f. PLoS One. 2013;8(2):e58004. doi: 10.1371/journal.pone.0058004. Epub 2013 Feb 28. PMID 23469127
- [Result] He X, Wang X, Fang J, Zhao Z, Huang L, Guo H, Zheng X. Bletilla striata: Medicinal uses, phytochemistry and pharmacological activities. J Ethnopharmacol. 2017 Jan 4;195:20-38. doi: 10.1016/j.jep.2016.11.026. Epub 2016 Nov 16. PMID 27865796
- [Result] Xu D, Pan Y, Chen J. Chemical Constituents, Pharmacologic Properties, and Clinical Applications of Bletilla striata. Front Pharmacol. 2019 Nov 1;10:1168. doi: 10.3389/fphar.2019.01168. eCollection 2019. PMID 31736742
- [Result] Zhang RX, Li MX, Jia ZP. Rehmannia glutinosa: review of botany, chemistry and pharmacology. J Ethnopharmacol. 2008 May 8;117(2):199-214. doi: 10.1016/j.jep.2008.02.018. Epub 2008 Mar 10. PMID 18407446
- [Result] Lim DW, Kim YT. Dried root of Rehmannia glutinosa prevents bone loss in ovariectomized rats. Molecules. 2013 May 17;18(5):5804-13. doi: 10.3390/molecules18055804. PMID 23685937
- [Result] Feng JC, Cai ZL, Zhang XP, Chen YY, Chang XL, Wang XF, Qin CB, Yan X, Ma X, Zhang JX, Nie GX. The Effects of Oral Rehmannia glutinosa Polysaccharide Administration on Immune Responses, Antioxidant Activity and Resistance Against Aeromonas hydrophila in the Common Carp, Cyprinus carpio L. Front Immunol. 2020 May 8;11:904. doi: 10.3389/fimmu.2020.00904. eCollection 2020. PMID 32457762
- [Result] Li HW, Liu P, Zhang HQ, Feng WM, Yan H, Guo S, Qian DW, Duan JA. Determination of bioactive compounds in the nonmedicinal parts of Scrophularia ningpoensis using ultra-high-performance liquid chromatography coupled with tandem mass spectrometry and chemometric analysis. J Sep Sci. 2020 Nov;43(22):4191-4201. doi: 10.1002/jssc.202000723. Epub 2020 Oct 12. PMID 32975375
- [Result] Ren D, Shen ZY, Qin LP, Zhu B. Pharmacology, phytochemistry, and traditional uses of Scrophularia ningpoensis Hemsl. J Ethnopharmacol. 2021 Apr 6;269:113688. doi: 10.1016/j.jep.2020.113688. Epub 2020 Dec 16. PMID 33338592
- [Result] Wang J, Huang L, Ren Q, Wang Y, Zhou L, Fu Y, Sai C, Pella SS, Guo Y, Gao LN. Polysaccharides of Scrophularia ningpoensis Hemsl.: Extraction, Antioxidant, and Anti-Inflammatory Evaluation. Evid Based Complement Alternat Med. 2020 Dec 15;2020:8899762. doi: 10.1155/2020/8899762. eCollection 2020. PMID 33381217
- [Result] Wang Z, He C, Peng Y, Chen F, Xiao P. Origins, Phytochemistry, Pharmacology, Analytical Methods and Safety of Cortex Moutan (Paeonia suffruticosa Andrew): A Systematic Review. Molecules. 2017 Jun 7;22(6):946. doi: 10.3390/molecules22060946. PMID 28590441
- [Result] Zhang L, Li DC, Liu LF. Paeonol: pharmacological effects and mechanisms of action. Int Immunopharmacol. 2019 Jul;72:413-421. doi: 10.1016/j.intimp.2019.04.033. Epub 2019 Apr 25. PMID 31030097
- [Result] Li P, Shen J, Wang Z, Liu S, Liu Q, Li Y, He C, Xiao P. Genus Paeonia: A comprehensive review on traditional uses, phytochemistry, pharmacological activities, clinical application, and toxicology. J Ethnopharmacol. 2021 Apr 6;269:113708. doi: 10.1016/j.jep.2020.113708. Epub 2020 Dec 24. PMID 33346027
- [Result] Stasiak N, Kukula-Koch W, Glowniak K. Modern industrial and pharmacological applications of indigo dye and its derivatives--a review. Acta Pol Pharm. 2014 Mar-Apr;71(2):215-21. PMID 25272640
- [Result] Qi-Yue Y, Ting Z, Ya-Nan H, Sheng-Jie H, Xuan D, Li H, Chun-Guang X. From natural dye to herbal medicine: a systematic review of chemical constituents, pharmacological effects and clinical applications of indigo naturalis. Chin Med. 2020 Dec 14;15(1):127. doi: 10.1186/s13020-020-00406-x. PMID 33317592
- [Result] Gu S, Xue Y, Gao Y, Shen S, Zhang Y, Chen K, Xue S, Pan J, Tang Y, Zhu H, Wu H, Dou D. Mechanisms of indigo naturalis on treating ulcerative colitis explored by GEO gene chips combined with network pharmacology and molecular docking. Sci Rep. 2020 Sep 16;10(1):15204. doi: 10.1038/s41598-020-71030-w. PMID 32938944
- [Result] El-Saber Batiha G, Magdy Beshbishy A, El-Mleeh A, Abdel-Daim MM, Prasad Devkota H. Traditional Uses, Bioactive Chemical Constituents, and Pharmacological and Toxicological Activities of Glycyrrhiza glabra L. (Fabaceae). Biomolecules. 2020 Feb 25;10(3):352. doi: 10.3390/biom10030352. PMID 32106571
- [Result] Pastorino G, Cornara L, Soares S, Rodrigues F, Oliveira MBPP. Liquorice (Glycyrrhiza glabra): A phytochemical and pharmacological review. Phytother Res. 2018 Dec;32(12):2323-2339. doi: 10.1002/ptr.6178. Epub 2018 Aug 17. PMID 30117204
- [Result] Isbrucker RA, Burdock GA. Risk and safety assessment on the consumption of Licorice root (Glycyrrhiza sp.), its extract and powder as a food ingredient, with emphasis on the pharmacology and toxicology of glycyrrhizin. Regul Toxicol Pharmacol. 2006 Dec;46(3):167-92. doi: 10.1016/j.yrtph.2006.06.002. Epub 2006 Aug 1. PMID 16884839
- [Result] Mangal P, Khare P, Jagtap S, Bishnoi M, Kondepudi KK, Bhutani KK. Screening of six Ayurvedic medicinal plants for anti-obesity potential: An investigation on bioactive constituents from Oroxylum indicum (L.) Kurz bark. J Ethnopharmacol. 2017 Feb 2;197:138-146. doi: 10.1016/j.jep.2016.07.070. Epub 2016 Jul 26. PMID 27469197
- [Result] Harminder, Singh V, Chaudhary AK. A Review on the Taxonomy, Ethnobotany, Chemistry and Pharmacology of Oroxylum indicum Vent. Indian J Pharm Sci. 2011 Sep;73(5):483-90. doi: 10.4103/0250-474X.98981. PMID 22923859
- [Result] Chen J, Chen J, Lu J. Systematic Elucidation of the Mechanism of Oroxylum indicum via Network Pharmacology. Evid Based Complement Alternat Med. 2020 Jul 14;2020:5354215. doi: 10.1155/2020/5354215. eCollection 2020. PMID 32733583